CLINICAL TRIAL: NCT02700724
Title: Observation Versus Immediate Surgery of Low Risk Bladder Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: poor enrollment
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Daniel Lee, Instructor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 151898
Record Dates: First submitted 2015-12-07; First posted 2016-03-07 (Estimated); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Transurethral Resection of Bladder; Observation; Watchful Waiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Observation (Other): Patients will not undergo immediate surgery. These patients will undergo surveillance cystoscopy and urinary cytology every 3 months for 12 months. Surgery will commence after 12 months of observation or sooner if cystoscopic evidence of disease progression or patient desire.
  Interventions: Other: Observation; Procedure: Surveillance Cystoscopy and Urinary Cytology
- Immediate Surgery (Other): Patients will undergo immediate surgery. These patients will undergo surveillance cystoscopy and urinary cytology every 3 months for 12 months. Repeated surgery will be offered for additional recurrences.
  Interventions: Other: Immediate Surgery; Procedure: Surveillance Cystoscopy and Urinary Cytology

INTERVENTIONS:
Other: Immediate Surgery
  Other Names: Transurethral Resection of Bladder Tumor
  Arms: Immediate Surgery
Other: Observation
  Other Names: Active Surveillance
  Arms: Observation
Procedure: Surveillance Cystoscopy and Urinary Cytology — Cytology and cystoscopy are done at the same time

SUMMARY:
This trial is a randomized, multi-center, non-inferiority study comparing observation versus immediate surgery for low grade, noninvasive bladder cancer.

ELIGIBILITY:
Inclusion Criteria:

* History of low grade, noninvasive urothelial carcinoma of the bladder with a new recurrence that meets the following criteria:
* total tumor burden ≤3cm in size (multiple lesions permitted)
* low grade appearance (grade 1 or grade 2)
* noninvasive appearance (Ta)
* no history of carcinoma in situ (CIS) or lesions concerning for CIS
* negative urine cytology (atypical or suspicious for low grade neoplasm are acceptable)

Exclusion Criteria:

* High grade and/or invasive and/or carcinoma in situ disease
* Concomitant upper tract urothelial carcinoma
* Any patient who is pregnant or who may have plans to become pregnant.
* Positive cytology

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-04; Primary Completion 2018-07-19 (Actual); Study Completion 2018-07-19 (Actual)

PRIMARY OUTCOMES:
Event-Free Survival | 12 months
  An event is a complication of any kind, including bleeding requiring blood transfusion, bladder perforation, urinary tract infection, readmission to the hospital, and progression of disease.

SECONDARY OUTCOMES:
Proportion of patients with disease progression (either stage or grade) | 12 months
  proportion of patients with disease progression (either stage or grade)
Patient-reported Costs | At baseline and 3 months, 6 months, 9 months and 12 months.
  out of pocket medical costs
Self-reported patient anxiety measured using the EORTC QLQ-NMIBC24 | At baseline and 3 months, 6 months, 9 months and 12 months.
  Measured using the EORTC QLQ-NMIBC24, which is a 24-item questionnaire for patients with superficial bladder cancer. This will be assessed at baseline and every 3 months during the study.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel D. Lee, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States